CLINICAL TRIAL: NCT06015113
Title: Efficacy and Safety of Disitamab Vedotin Plus Pyrotinib or Naratinib in HER2-positive Breast Cancer Patients With Brain Metastasis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xi'an International Medical Center Hospital (Other)
Responsible Party: Principal Investigator, Yan Xue, Director of tumor hospital, Xi'an International Medical Center Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECCO-KY-22004
Record Dates: First submitted 2023-08-08; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — disitamab vedotin; pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Label 1 (Experimental): tale Disitamab Vedotin with pyrotinib or neratinib
  Interventions: Drug: Disitamab Vedotin plus pyrotinib or naratinib

INTERVENTIONS:
Drug: Disitamab Vedotin plus pyrotinib or naratinib — Trastuzumab Injection: Intravenous infusion, initial loading dose of 2 mg/kg, administered via intravenous infusion over 30-90 minutes (usually recommended around 60 minutes), administered on day 1 of each cycle, with each cycle lasting 14 days.
  Pyrotinib Maleate Tablets: 400 mg, taken orally once daily, within 30 minutes after a meal, at the same time every day. Taken continuously, with each cycle lasting 14 days.
  Neratinib Maleate Tablets: 240 mg, taken orally once daily with a meal, at the same time every day. The neratinib tablet should be swallowed whole (it should not be chewed, crushed, or split before swallowing). Taken continuously, with each cycle lasting 14 days.

SUMMARY:
Basis: Brain metastasis is very common in breast cancer, and HER2 positivity is a risk factor for high incidence of brain metastasis, with approximately 50% of HER2+ MBC cases experiencing brain metastasis. The reason for this is that as the efficacy of HER2-targeted therapy improves, the survival of these patients significantly extends, leading to an increase in the occurrence rate of brain metastasis events in the late stage of MBC. In the systemic treatment of HER2+ breast cancer brain metastasis, various HER2-targeted drugs have been explored, but none have achieved satisfactory therapeutic effects. Therefore, it is imperative to explore new treatment options. ADC drugs have shown some efficacy in brain metastasis patients, and as a domestically developed ADC drug, trastuzumab vedotin has demonstrated good anti-tumor effects. The treatment model combining trastuzumab vedotin with small molecule TKIs has been rarely reported, so we are attempting to use the treatment model of trastuzumab vedotin combined with pyrotinib or neratinib to explore its efficacy and safety in patients with HER2-positive brain metastasis.

Method: The plan is to recruit HER2-positive breast cancer patients with brain metastasis and use the treatment of trastuzumab vedotin combined with pyrotinib or neratinib (specific treatment drugs to be selected during the study).

Procedure: All subjects will undergo screening, treatment, and follow-up periods, strictly adhering to relevant GCP regulations during the treatment process.

Expectations: Through this study, preliminary efficacy and safety data of trastuzumab vedotin combined with pyrotinib or neratinib treatment will be provided for patients with HER2+ brain metastatic BC.

DETAILED DESCRIPTION:
Treatment Plan After patient screening, patients will receive treatment with trastuzumab injection plus either pyrotinib maleate tablets or neratinib maleate tablets, with each cycle lasting 14 days until disease progression. Trastuzumab Injection: Intravenous infusion, initial loading dose of 2 mg/kg, administered via intravenous infusion over 30-90 minutes (usually recommended around 60 minutes), administered on day 1 of each cycle, with each cycle lasting 14 days. Pyrotinib Maleate Tablets: 400 mg, taken orally once daily, within 30 minutes after a meal, at the same time every day. Taken continuously, with each cycle lasting 14 days. If a patient misses a dose of pyrotinib, it should not be made up for, and the next dose should be taken as scheduled. Neratinib Maleate Tablets: 240 mg, taken orally once daily with a meal, at the same time every day. The neratinib tablet should be swallowed whole (it should not be chewed, crushed, or split before swallowing). Taken continuously, with each cycle lasting 14 days. If a patient misses a dose of neratinib, it should not be made up for, and the next dose should be taken as scheduled. Note: The choice between pyrotinib maleate tablets or neratinib maleate tablets for treatment should be based on the patient's previous treatment history as decided by the investigator. Treatment medication should be continued until disease progression or the occurrence of intolerable toxic reactions.

Study Steps 1) Screening Period (Visit 1: -14 to -1 days, approximately 2 weeks): Subjects will sign an informed consent form during Visit 1 and undergo a series of examinations (see Table 1. Treatment Flowchart). Based on the examination results and inclusion/exclusion criteria, the investigator will determine if the subject meets the inclusion criteria and does not meet the exclusion criteria. 2) Treatment Period (Visit 2 to disease progression, 1 visit every 2 cycles): Subjects will receive treatment with trastuzumab injection plus pyrotinib maleate tablets plus capecitabine tablets on the experimental Day 0, with each cycle lasting 21 days, until disease progression. During this period, a series of examinations will be conducted every 2 cycles (see flowchart for visits 2 to N). The investigator will evaluate the effectiveness and safety of the treatment based on the subject's examination results. 3) Survival Follow-up Period (1 follow-up every 3 months after withdrawal from the study): After patients withdraw due to disease progression or other endpoint events, a telephone follow-up will be conducted every 3 months until the patient's death or loss to follow-up. Detailed records of disease progression, related treatments, and survival information should be documented.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can voluntarily sign an informed consent form;
* Females aged ≥18 years old when signing the informed consent form;
* ECOG PS physical status score of 0 to 2 points;
* Histologically confirmed HER2-positive metastatic breast cancer patients; Note: HER2 positivity refers to at least one occurrence of tumor cell immunohistochemical staining intensity of 3+ or confirmed as positive by fluorescence in situ hybridization [FISH] in the pathological testing/re-review of the primary or metastatic lesions conducted by the participating center's pathology department;
* Brain metastases confirmed by MRI/enhanced CT, with at least one measurable lesion in the brain based on RECIST 1.1 criteria;
* Expected survival period ≥3 months;
* Patient types: Cohort A - newly diagnosed brain metastases patients; Cohort B - patients with progression after whole-brain radiotherapy or stereotactic radiosurgery;
* Left ventricular ejection fraction (LVEF) ≥50%;
* QT interval corrected by Fridericia formula (QTcF) of 12-lead electrocardiogram: <450ms for males, <470ms for females;
* The following conditions should be met in the blood routine examination:① Absolute neutrophil count (ANC) ≥1.5×10^9/L, ② Platelet count ≥100×10^9/L, ③ Hemoglobin ≥90g/L, ④ White blood cell count ≥3.0×10^9/L;
* Liver function meets the following conditions: ① Serum total bilirubin ≤1.5×upper limit of normal (ULN), or ≤3×ULN if there are liver metastases, ② Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤3×ULN, or ≤5×ULN if there are liver metastases;
* Renal function meets the following conditions: Serum creatinine ≤1.5×ULN or creatinine clearance ≥50mL/min (calculated according to the Cockroft-Gault formula);
* Female patients who meet the following conditions can participate in this study: ① Infertility; ② Capable of fertility, with a negative blood pregnancy test result within 7 days before the first administration of the investigational drug, not breastfeeding, and adopting effective contraceptive measures during the screening period, throughout the study, and within 6 months after the last administration of the study drug.

Exclusion Criteria:

* Patients who have received treatment with anti-HER2 ADC drugs;
* Patients who have received sequential treatment with pyrotinib and neratinib;
* Patients with extensive leptomeningeal metastases and poor response to steroid dehydration therapy for brain metastases;
* Presence of third space fluid accumulation (such as significant pleural effusion or ascites) that cannot be controlled by drainage or other methods;
* Patients who have received chemotherapy, major surgery, or molecular targeted therapy within 2 weeks prior to enrollment; patients who have received endocrine therapy within 1 week prior to enrollment; patients who have received nitrosoureas or mitomycin chemotherapy within 6 weeks prior to enrollment;
* Concurrent use of any other anticancer treatment;
* History of or current concurrent malignancies within the past 5 years, excluding cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder carcinoma [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor invading the lamina propria)];
* Underwent major surgery (including thoracotomy biopsy), experienced significant trauma (such as fractures), had unhealed wounds or fractures at the time of screening, or anticipated the need for major surgery during the study treatment period, within the 4 weeks prior to randomization;
* History of myocardial infarction within the past 6 months; history of New York Heart Association (NYHA) class ≥II congestive heart failure that is not controlled by medication, severe arrhythmias that cannot be controlled (excluding atrial fibrillation and paroxysmal supraventricular tachycardia); known decrease in LVEF to below 50% during or after previous treatment with trastuzumab;
* Known allergy to the drugs and excipients involved in this trial;
* Known history of hypersensitivity reactions to any investigational drugs;
* Subjects deemed unsuitable for participation by other investigators.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | The time from randomization to the first documented tumor progression or death from any cause, whichever came first, assessed up to 100 months
  It is an indicator of the long-term efficacy of the drug.

SECONDARY OUTCOMES:
Objective Response Rate | 4 weeks
  The proportion of patients with the best response of complete response (CR) or partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST).
Disease Control Rate | 4 weeks
  The proportion of patients with tumor shrinkage or stability maintained for a certain period, including cases of CR, PR, and stable disease (SD)
Overall survival | the time from randomization to death from any cause，whichever came first, assessed up to 100 months.
  It is an indicator of the long-term efficacy of the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Xue, Principal Investigator — Xi'an International Medical Center Hospital
Locations (1):
- Xi'an International Medical Center Hospital, Xi'an, Shaanxi, China